CLINICAL TRIAL: NCT05107557
Title: A Randomized and Controlled Phase IV Clinical Trial to Evaluate the Immunogenicity and Safety of COVID-19 Vaccine (Vero Cell), Inactivated Co-administrated With EV71 Vaccine (Vero Cell) in Children Aged 3-5 Years Old
Brief Title: Immunogenicity And Safety of COVID-19 Vaccine , Inactivated Co -Administration With EV71 Vaccine (Vero Cell)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-4002-1
Record Dates: First submitted 2021-11-02; First posted 2021-11-04 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group is also called the combined immunization group.260 participants will receive the first dose of COVID-19 vaccine and EV71 vaccine on day 0 and the second dose of COVID-19 vaccine and EV71 vaccine on day 28.
  Interventions: Biological: Experimental Group
- Control Group (Active Comparator): The control group is also called the Non-combined immunization group.260 participants will receive the first dose of COVID-19 vaccine on day 0,the first dose of EV71 vaccine on day 14,the second dose of COVID-19 vaccine on day 28 and the second dose of EV71 vaccine on day 42.
  Interventions: Biological: Experimental Group

INTERVENTIONS:
Biological: Experimental Group — The COVID-19 vaccine was manufactured by Sinovac Research & Development Co., Ltd, and the EV71 vaccine was manufactured by Sinovac Biotech Co.The COVID-19 vaccine:600SU inactivated virus in 0.5mL of aluminium hydroxide solution per injection;The EV71 vaccine:Inactivated EV71 virus antigen no less than 3.0EU in 0.5 mL of aluminium hydroxide solution per injection.
  Other Names: Combined immunization group

SUMMARY:
This study is a randomized and controlled Phase IV clinical trial of the COVID-19 vaccine (Vero cell), Inactivated manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the immunogenicity and safety of COVID-19 vaccine (Vero cell), Inactivated co-administration with EV71 vaccine

DETAILED DESCRIPTION:
This study is a randomized and controlled phase IV clinical trial in children aged 3-5 years old. The purpose of this study is to evaluate the immunogenicity and safety of COVID-19 vaccine (Vero cell), Inactivated co-administration with EV71 vaccine.The COVID-19 vaccine was manufactured by Sinovac Research & Development Co., Ltd and the EV71 vaccine was manufactured by Sinovac Biotech Co.A total of 520 subjects aged 3-5 years old will be enrolled.Subjects will be randomly divided into 2 groups in a ratio of 1:1.The experimental group is the combined immunization group, which will receive the first dose of COVID-19 vaccine and the first dose of EV71 vaccine on day 0 and the second dose of COVID-19 vaccine and EV71 vaccine on day 28;Control group is the Non-combined immunization group , which will receive the first dose of COVID-19 vaccine on day 0 ,the first dose of EV71 vaccine on day 14, the second dose of COVID-19 vaccine on day 28 and the second dose of EV71 vaccine on day 42.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-5 years;
* The subject and/or guardian can understand and voluntarily sign the informed consent form;
* Proven legal identity.

Exclusion Criteria:

* History of contact with a SARS-CoV-2 infection (positive in nucleic acid test) within 14 days;
* History of multiple system inflammatory syndrome (MIS-C);
* History of hand, foot and mouth disease, herpetic angina or EV71 vaccination;
* History of asthma, history of allergy to the vaccine or vaccine components,or serious adverse reactions to the vaccine, such as urticaria, dyspnea,and angioedema;
* Congenital malformations or developmental disorders, genetic defects,severe malnutrition, etc.;
* Autoimmune disease (Systemic lupus erythematosus)or immunodeficiency / immunosuppression(HIV,history after organ transplantation);
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases,malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, asplenia,functional asplenia, asplenia or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy,abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Axillary temperature >37.0°C;
* The subjects participated in other clinical trials during the follow-up period,or will be planned within 3 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index-Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 | Day 28 after the second dose of COVID-19 vaccine
  Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose of COVID-19 vaccine
Immunogenicity index-Seroconversion rate of the neutralizing antibody to EV71 | Day 28 after the second dose of EV71 vaccine
  Seroconversion rate of the neutralizing antibody to EV71 at day 28 after the second dose of EV71 vaccine

SECONDARY OUTCOMES:
Immunogenicity index-Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 | Day 28 after the second dose of COVID-19 vaccine
  Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose of COVID-19 vaccine.
Immunogenicity index- GMT of the neutralizing antibody to live SARS-CoV-2 | Day 28 after the second dose of COVID-19 vaccine
  GMT of the neutralizing antibody to live SARS-CoV-2 at day 28 after after the second dose of COVID-19 vaccine.
Immunogenicity index-GMI of the neutralizing antibody to live SARS-CoV-2 | Day 28 after the second dose of COVID-19 vaccine
  GMI of the neutralizing antibody to live SARS-CoV-2 at day 28 after after the second dose of COVID-19 vaccine.
Immunogenicity index-Seropositive rate of the neutralizing antibody to EV71 | Day 28 after the second dose of EV71
  Seropositive rate of the neutralizing antibody to EV71 at day 28 after the second dose of EV71
Immunogenicity index-GMT of the neutralizing antibody to EV71 | Day 28 after the second dose of EV71
  GMT of the neutralizing antibody to EV71 at day 28 after the second dose of EV71
Immunogenicity index-GMI of the neutralizing antibody to EV71 | Day 28 after the second dose of EV71
  GMI of the neutralizing antibody to EV71 at day 28 after the second dose of EV71
Safety index-Incidence of the adverse reactions | From day 0 to day 7 after each dose
  Incidence of the adverse reactions from day 0 to day 7 after each dose
Safety index-Incidence of the adverse reactions | From day 0 to 28 days after the last dose
  Incidence of the adverse reactions from day 0 to 28 days after the last dose
Safety index-Incidence of the serious adverse events and the adverse events of special concern | From the beginning vaccination to 6 months after the last dose
  Incidence of the serious adverse events and the adverse events of special concern from the beginning vaccination to 6 months after the last dose

OTHER OUTCOMES:
Immunogenicity index-Seropositive rate of the neutralizing antibody to live SARS-CoV-2 | 6 months after the second dose of COVID-19 vaccine
  Seropositive rate and GMT of the neutralizing antibody to live SARS-CoV-2 6 months after the second dose of COVID-19 vaccine
Immunogenicity index- GMT of the neutralizing antibody to live SARS-CoV-2 | 6 months after the second dose of COVID-19 vaccine
  GMT of the neutralizing antibody to live SARS-CoV-2 6 months after the second dose of COVID-19 vaccine
Immunogenicity index-Seropositive rate of the neutralizing antibody to EV71 | 6 months after the second dose of EV71 vaccine
  Seropositive rate of the neutralizing antibody to EV71 6 months after the second dose of EV71 vaccine
Immunogenicity index-GMT of the neutralizing antibody to EV71 | 6 months after the second dose of EV71 vaccine
  GMT of the neutralizing antibody to EV71 6 months after the second dose of EV71 vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuhang Huang, Master, Principal Investigator — Guangdong Center for Disease Prevention and Control
Locations (2):
- China (2):
  - Yangchun City Center for Disease Control and Prevention, Yangchun, Guangdong
  - Zhanjiang Center for Diseases Control and Prevention, Zhenjiang, Guangdong